CLINICAL TRIAL: NCT01473043
Title: Clinical Study With Axitinib (AG 013736) In Patients With Metastatic Renal Cell Carcinoma After Failure Of One Prior Systemic First-Line Therapy
Brief Title: Clinical Study With Axitinib In Advanced Kidney Cancer, Who Have Failed First Line Treatment
Status: No longer available | Type: Expanded Access
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A4061061
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Renal Cell Carcinoma
Keywords: Axitinib; metastatic renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Axitinib

INTERVENTIONS:
Drug: Axitinib — 5mg twice daily [BD] daily dosing until progression or prohibitive toxicity Dose titration by 2 levels upwards (7mg and 10mg) and downwards (3mg and 2mg) allowed per protocol
  Other Names: AG-013736

SUMMARY:
This is a single arm study with axitinib in patients with advanced kidney cancer (clear cell variant), who have failed first line therapy. The study will recruit a maximum of 30 patients from 2 countries including Australia and Canada. Patients will be followed up for efficacy, safety and health related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic renal cell carcinoma with a component of clear cell subtype.
* Prior first line systemic therapy
* At least 1 measurable lesion as per Response Evaluation Criterion in Solid Tumors [RECIST 1.1].
* Adequate hematology, liver and kidney functions
* Eastern Cooperative Oncology Group [ECOG] performance status of 0 or 1.
* Life expectancy of ≥12 weeks.
* Normotensive or well controlled hypertension (less than/equal to 140/90 mm Hg.)
* Negative pregnancy test
* Adequate recovery time from prior systemic therapy, surgery or radiation
* Willing and able subjects who have signed consent

Exclusion Criteria:

* More than one prior systemic therapy regimen
* Major bowel-penetrating surgery <4 weeks
* Active gastro intestinal bleed in past 3 months
* Active peptic ulcer disease in the past 6 months
* Current or anticipated use of potent CYP3A4/5 inhibitors
* Current or anticipated use of known CYP3A4/5 or CYP1A2 inducers
* Requirement for therapeutic warfarin or high dose steroids
* Symptomatic or untreated brain metastases
* A serious uncontrolled medical disorder or active infection
* Pregnant or breastfeeding females
* History of another active malignancy
* Dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2012-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Australia (3):
  - Pfizer Investigational Site, Douglas, Queensland
  - Pfizer Investigational Site, Hobart, Tasmania
  - Pfizer Investigational Site, Wendouree, Victoria
- Pfizer Investigational Site, Montreal, Quebec, Canada

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061061&StudyName=Clinical%20Study%20With%20Axitinib%20In%20Advanced%20Kidney%20Cancer%2C%20Who%20Have%20Failed%20First%20Line%20Treatment%20